CLINICAL TRIAL: NCT03641651
Title: Feasibility and Cost Description of Intensive Rehabilitation Involving New Technologies in Patients With Sub-acute Stroke:A Multicenter Single Arm Trial of the Swiss RehabTech Initiative
Brief Title: New Technologies in the Rehabilitation of Chronic Stroke
Acronym: SRTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Markus Wirz (Other)
Collaborators: Klinik Lengg, Zurich (Other); Reha Rheinfelden (Other); Klinik Valens (Other); Rehaklinik Zihlschlacht AG (Other)
Responsible Party: Sponsor-Investigator, Markus Wirz, Head of Physiotherapy R&D, Zurich University of Applied Sciences
Organization: Zurich University of Applied Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ZHAW-SRTI
Record Dates: First submitted 2018-08-13; First posted 2018-08-22 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Stroke; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — frovatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Technology arm (Experimental): 4 Weeks intervention of intensive rehabilitation using rehabilitation technology, 3-5 h per day, within a 5d week in-or outpatient setting.
  Interventions: Other: Rehabilitation technology

INTERVENTIONS:
Other: Rehabilitation technology — * Series of tailored rehabilitative training with the use of new technology which provide feedback and allow for a targeted and intensive and dense training.
  * With supervision based on patients preconditions and therapy device (e.g. patient/ therapist ratio= 3/1).
  * A training series lasts four weeks and comprises 3-5 training-days per week. Maximum training break of 7 days.
  Five sessions of training with duration of 45 min per session, and up to four hours each day are foreseen.
  * The training can take place in an outpatient or inpatient setting.
  * Training will be organized in individual one-to-one or group session
  Other Names: Lokomat; Erigo; Andago; Armeo (Boom, Senseo, Spring, Power); Valedo motion; Amadeo; Myro; NuStep; Bi-Manu Trainer; EksoGT; The Float; MOTOmed; Allegro

SUMMARY:
The objective of the current study is to develop and investigate training concepts involving rehabilitation technology, which aim at exploiting the potential for regaining the ability to perform skilled movements by maximizing training intensity and keeping the motivation of patients high.

The evaluation focuses on feasibility and cost-benefit analyses

DETAILED DESCRIPTION:
This feasibility project aims to establish an efficient setting for intensive rehabilitation with new technology in four trailblazer clinics. This will enable them to provide intensive therapy to the patients in accordance with the study protocol. If this setting is integrated into the clinical routine, the investigators will be able to collect data to get some first insight into economic and functional data required to calculate changes in socioeconomic costs

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with residual hemiparesis after cerebrovascular accident
* Up to 12 months after the event
* Primary rehabilitation terminated
* Able to cognitively comprehend the aim of the project with at least 22 points in the Montreal Cognitive Assessment (MoCA)
* General health condition allows for intensive rehabilitative training with limited supervision i.e. clearance and prescription of responsible physician
* Understand written and spoken German language

Exclusion Criteria:

Patients with any signs and symptoms showing that the participant is unwilling to participate in the study will result in the patient being excluded from participation Any medical condition preventing participation such as Severe respiratory disease Severe OR unstable cardio-circulatory conditions Orthopaedic conditions, especially in extremities targeted for rehabilitation such as

* fixed joint contractures limiting range of motion
* non-consolidated fractures Neuro-psychological conditions including cognitive deficits limiting communication or non-cooperation like (self-) aggressive behaviour Infections or inflammatory diseases, like osteomyelitis

Specific absolute contraindication for the training with any of the respective devices:

* Improper fit of the device, including its harness to relevant extremity(ies)
* Contraindicated training position (standing, sitting)

Device specific contraindications will be respected and will lead to the exclusion of the device for that patient.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Switzerland (4):
  - Reha Rheinfelden, Rheinfelden
  - Kliniken Valens, Valens
  - Rehakliniken Zihlschlacht, Zihlschlacht
  - Klinik Lengg AG, Zurich

REFERENCES:
- [Background] Pollock A, Baer G, Campbell P, Choo PL, Forster A, Morris J, Pomeroy VM, Langhorne P. Physical rehabilitation approaches for the recovery of function and mobility following stroke. Cochrane Database Syst Rev. 2014 Apr 22;2014(4):CD001920. doi: 10.1002/14651858.CD001920.pub3. PMID 24756870
- [Background] Veerbeek JM, van Wegen E, van Peppen R, van der Wees PJ, Hendriks E, Rietberg M, Kwakkel G. What is the evidence for physical therapy poststroke? A systematic review and meta-analysis. PLoS One. 2014 Feb 4;9(2):e87987. doi: 10.1371/journal.pone.0087987. eCollection 2014. PMID 24505342
- [Background] Langhorne P, Wagenaar R, Partridge C. Physiotherapy after stroke: more is better? Physiother Res Int. 1996;1(2):75-88. doi: 10.1002/pri.6120010204. PMID 9238725
- [Background] Hornby TG, Holleran CL, Hennessy PW, Leddy AL, Connolly M, Camardo J, Woodward J, Mahtani G, Lovell L, Roth EJ. Variable Intensive Early Walking Poststroke (VIEWS): A Randomized Controlled Trial. Neurorehabil Neural Repair. 2016 Jun;30(5):440-50. doi: 10.1177/1545968315604396. Epub 2015 Sep 3. PMID 26338433
- [Background] Knecht S, Rossmuller J, Unrath M, Stephan KM, Berger K, Studer B. Old benefit as much as young patients with stroke from high-intensity neurorehabilitation: cohort analysis. J Neurol Neurosurg Psychiatry. 2016 May;87(5):526-30. doi: 10.1136/jnnp-2015-310344. Epub 2015 Jun 11. PMID 26069298
- [Background] Kwakkel G, Wagenaar RC, Twisk JW, Lankhorst GJ, Koetsier JC. Intensity of leg and arm training after primary middle-cerebral-artery stroke: a randomised trial. Lancet. 1999 Jul 17;354(9174):191-6. doi: 10.1016/S0140-6736(98)09477-X. PMID 10421300
- [Background] Feys H, De Weerdt W, Verbeke G, Steck GC, Capiau C, Kiekens C, Dejaeger E, Van Hoydonck G, Vermeersch G, Cras P. Early and repetitive stimulation of the arm can substantially improve the long-term outcome after stroke: a 5-year follow-up study of a randomized trial. Stroke. 2004 Apr;35(4):924-9. doi: 10.1161/01.STR.0000121645.44752.f7. Epub 2004 Mar 4. PMID 15001789
- [Background] Jette DU, Warren RL, Wirtalla C. The relation between therapy intensity and outcomes of rehabilitation in skilled nursing facilities. Arch Phys Med Rehabil. 2005 Mar;86(3):373-9. doi: 10.1016/j.apmr.2004.10.018. PMID 15759214
- [Background] Lohse KR, Lang CE, Boyd LA. Is more better? Using metadata to explore dose-response relationships in stroke rehabilitation. Stroke. 2014 Jul;45(7):2053-8. doi: 10.1161/STROKEAHA.114.004695. Epub 2014 May 27. PMID 24867924
- [Background] Birkenmeier RL, Prager EM, Lang CE. Translating animal doses of task-specific training to people with chronic stroke in 1-hour therapy sessions: a proof-of-concept study. Neurorehabil Neural Repair. 2010 Sep;24(7):620-35. doi: 10.1177/1545968310361957. Epub 2010 Apr 27. PMID 20424192
- [Background] Kwakkel G, van Peppen R, Wagenaar RC, Wood Dauphinee S, Richards C, Ashburn A, Miller K, Lincoln N, Partridge C, Wellwood I, Langhorne P. Effects of augmented exercise therapy time after stroke: a meta-analysis. Stroke. 2004 Nov;35(11):2529-39. doi: 10.1161/01.STR.0000143153.76460.7d. Epub 2004 Oct 7. PMID 15472114
- [Background] Teasell R, Bitensky J, Salter K, Bayona NA. The role of timing and intensity of rehabilitation therapies. Top Stroke Rehabil. 2005 Summer;12(3):46-57. doi: 10.1310/ETDP-6DR4-D617-VMVF. PMID 16110427
- [Background] Andrews AW, Li D, Freburger JK. Association of Rehabilitation Intensity for Stroke and Risk of Hospital Readmission. Phys Ther. 2015 Dec;95(12):1660-7. doi: 10.2522/ptj.20140610. Epub 2015 Jun 18. PMID 26089042
- [Background] Krakauer JW, Carmichael ST, Corbett D, Wittenberg GF. Getting neurorehabilitation right: what can be learned from animal models? Neurorehabil Neural Repair. 2012 Oct;26(8):923-31. doi: 10.1177/1545968312440745. Epub 2012 Mar 30. PMID 22466792
- [Background] De Wit L, Putman K, Dejaeger E, Baert I, Berman P, Bogaerts K, Brinkmann N, Connell L, Feys H, Jenni W, Kaske C, Lesaffre E, Leys M, Lincoln N, Louckx F, Schuback B, Schupp W, Smith B, De Weerdt W. Use of time by stroke patients: a comparison of four European rehabilitation centers. Stroke. 2005 Sep;36(9):1977-83. doi: 10.1161/01.STR.0000177871.59003.e3. Epub 2005 Aug 4. PMID 16081860
- [Background] De Wit L, Putman K, Schuback B, Komarek A, Angst F, Baert I, Berman P, Bogaerts K, Brinkmann N, Connell L, Dejaeger E, Feys H, Jenni W, Kaske C, Lesaffre E, Leys M, Lincoln N, Louckx F, Schupp W, Smith B, De Weerdt W. Motor and functional recovery after stroke: a comparison of 4 European rehabilitation centers. Stroke. 2007 Jul;38(7):2101-7. doi: 10.1161/STROKEAHA.107.482869. Epub 2007 May 31. PMID 17540968
- [Background] Hayward KS, Brauer SG. Dose of arm activity training during acute and subacute rehabilitation post stroke: a systematic review of the literature. Clin Rehabil. 2015 Dec;29(12):1234-43. doi: 10.1177/0269215514565395. Epub 2015 Jan 7. PMID 25568073
- [Background] Lang CE, Macdonald JR, Reisman DS, Boyd L, Jacobson Kimberley T, Schindler-Ivens SM, Hornby TG, Ross SA, Scheets PL. Observation of amounts of movement practice provided during stroke rehabilitation. Arch Phys Med Rehabil. 2009 Oct;90(10):1692-8. doi: 10.1016/j.apmr.2009.04.005. PMID 19801058
- [Background] Lang CE, Wagner JM, Edwards DF, Dromerick AW. Upper extremity use in people with hemiparesis in the first few weeks after stroke. J Neurol Phys Ther. 2007 Jun;31(2):56-63. doi: 10.1097/NPT.0b013e31806748bd. PMID 17558358
- [Background] Taub E, Miller NE, Novack TA, Cook EW 3rd, Fleming WC, Nepomuceno CS, Connell JS, Crago JE. Technique to improve chronic motor deficit after stroke. Arch Phys Med Rehabil. 1993 Apr;74(4):347-54. PMID 8466415
- [Background] Gresham GE, Fitzpatrick TE, Wolf PA, McNamara PM, Kannel WB, Dawber TR. Residual disability in survivors of stroke--the Framingham study. N Engl J Med. 1975 Nov 6;293(19):954-6. doi: 10.1056/NEJM197511062931903. PMID 1178004
- [Background] Johnson BH, Bonafede MM, Watson C. Short- and longer-term health-care resource utilization and costs associated with acute ischemic stroke. Clinicoecon Outcomes Res. 2016 Feb 23;8:53-61. doi: 10.2147/CEOR.S95662. eCollection 2016. PMID 26966382
- [Background] McGuire AJ, Raikou M, Whittle I, Christensen MC. Long-term mortality, morbidity and hospital care following intracerebral hemorrhage: an 11-year cohort study. Cerebrovasc Dis. 2007;23(2-3):221-8. doi: 10.1159/000097645. Epub 2006 Dec 1. PMID 17143007
- [Background] Taylor TN, Davis PH, Torner JC, Holmes J, Meyer JW, Jacobson MF. Lifetime cost of stroke in the United States. Stroke. 1996 Sep;27(9):1459-66. doi: 10.1161/01.str.27.9.1459. PMID 8784113
- [Background] Zhao Y, Condon J, Lawton P, He V, Cadilhac DA. Lifetime direct costs of stroke for indigenous patients adjusted for comorbidities. Neurology. 2016 Aug 2;87(5):458-65. doi: 10.1212/WNL.0000000000002908. Epub 2016 Jul 1. PMID 27371489
- [Background] Duret C, Hutin E, Lehenaff L, Gracies JM. Do all sub acute stroke patients benefit from robot-assisted therapy? A retrospective study. Restor Neurol Neurosci. 2015;33(1):57-65. doi: 10.3233/RNN-140418. PMID 25420902
- [Background] Lo AC, Guarino PD, Richards LG, Haselkorn JK, Wittenberg GF, Federman DG, Ringer RJ, Wagner TH, Krebs HI, Volpe BT, Bever CT Jr, Bravata DM, Duncan PW, Corn BH, Maffucci AD, Nadeau SE, Conroy SS, Powell JM, Huang GD, Peduzzi P. Robot-assisted therapy for long-term upper-limb impairment after stroke. N Engl J Med. 2010 May 13;362(19):1772-83. doi: 10.1056/NEJMoa0911341. Epub 2010 Apr 16. PMID 20400552
- [Background] Spiess MR, Jaramillo JP, Behrman AL, Teraoka JK, Patten C. Unexpected recovery after robotic locomotor training at physiologic stepping speed: a single-case design. Arch Phys Med Rehabil. 2012 Aug;93(8):1476-84. doi: 10.1016/j.apmr.2012.02.030. Epub 2012 Mar 23. PMID 22446153
- [Background] Chang WH, Kim YH. Robot-assisted Therapy in Stroke Rehabilitation. J Stroke. 2013 Sep;15(3):174-81. doi: 10.5853/jos.2013.15.3.174. Epub 2013 Sep 27. PMID 24396811
- [Background] Masiero S, Poli P, Rosati G, Zanotto D, Iosa M, Paolucci S, Morone G. The value of robotic systems in stroke rehabilitation. Expert Rev Med Devices. 2014 Mar;11(2):187-98. doi: 10.1586/17434440.2014.882766. Epub 2014 Jan 30. PMID 24479445
- [Background] Tefertiller C, Pharo B, Evans N, Winchester P. Efficacy of rehabilitation robotics for walking training in neurological disorders: a review. J Rehabil Res Dev. 2011;48(4):387-416. doi: 10.1682/jrrd.2010.04.0055. PMID 21674390
- [Background] Waldner A, Tomelleri C, Hesse S. Transfer of scientific concepts to clinical practice: recent robot-assisted training studies. Funct Neurol. 2009 Oct-Dec;24(4):173-7. PMID 20412721
- [Background] Babaiasl M, Mahdioun SH, Jaryani P, Yazdani M. A review of technological and clinical aspects of robot-aided rehabilitation of upper-extremity after stroke. Disabil Rehabil Assist Technol. 2016;11(4):263-80. doi: 10.3109/17483107.2014.1002539. Epub 2015 Jan 20. PMID 25600057
- [Background] Mehrholz J, Thomas S, Werner C, Kugler J, Pohl M, Elsner B. Electromechanical-Assisted Training for Walking After Stroke: A Major Update of the Evidence. Stroke. 2017 Jun 16:STROKEAHA.117.018018. doi: 10.1161/STROKEAHA.117.018018. Online ahead of print. No abstract available. PMID 28626059
- [Background] Schuster-Amft C, Kool J, Moller JC, Schweinfurther R, Ernst MJ, Reicherzer L, Ziller C, Schwab ME, Wieser S, Wirz M; SRTI study group. Feasibility and cost description of highly intensive rehabilitation involving new technologies in patients with post-acute stroke-a trial of the Swiss RehabTech Initiative. Pilot Feasibility Stud. 2022 Jul 5;8(1):139. doi: 10.1186/s40814-022-01086-0. PMID 35791026

RESULTS

PARTICIPANT FLOW:
Groups:
- Technology Arm: 4 Weeks intervention of intensive rehabilitation using rehabilitation technology, 3-5 h per day, within a 5d week in-or outpatient setting.
  Rehabilitation technology: •Series of tailored rehabilitative training with the use of new technology which provide feedback and allow for a targeted and intensive and dense training.
  * With supervision based on patients preconditions and therapy device (e.g. patient/ therapist ratio= 3/1).
  * A training series lasts four weeks and comprises 3-5 training-days per week. Maximum training break of 7 days.
  Five sessions of training with duration of 45 min per session, and up to four hours each day are foreseen.
  * The training can take place in an outpatient or inpatient setting.
  * Training will be organized in individual one-to-one or group session
Period: Overall Study
Arm/Group | Technology Arm
Started | 15
Completed | 14
Not Completed | 1
Not completed — organizational issues at one study site | 1

BASELINE CHARACTERISTICS:
Arm/Group | Technology Arm
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 14
Paretic side [Count of Participants; unit: Participants] — Left /Right side
  Participants
    Left side | 9
    Right side | 5
Montreal Cognitive assessment (MoCA) [Mean (Standard Deviation); unit: units on a scale] — 0-30 points on scale, more points meaning better cognitive function
  units on a scale | 24.9 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Scheduled and Performed Trainings
Description: Adherence was operationalized by correlating planned trainings with trainings which were carried out by the participants. Due to the small sample size Spearman's rank correlation was used.
Time Frame: 4 weeks
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Technology Arm
Number analyzed (Participants) | 14
correlation coefficient | 0.56 [0.50 to 0.61]

2. Secondary Outcome: Functional Independence Measurement (FIM) Generic Functional Performance
Description: observer based measurement of the subject performing basic functional tests, e.g. sitting-up from lying position, stand-up from sitting, walking, stair-climbing etc. Observer rate on a scale from 1 to 7 (1= totally dependent on aid, 7= totally independent) for each activity 18 items, that would led to a score from 18 (totally dependent) to 126 (totally independent)
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Technology Arm
Number analyzed (Participants) | 14
units on a scale
  pre-intervention | 102 (47.5)
  post-intervention | 104.5 (32.5)

3. Secondary Outcome: Stroke Impact Scale (SIS) Recovery
Description: Questionnaire to be completed by the patient, regarding different parts in daily life: 1. physical problems: 4 items, 2. memory and thinking: 7 items, 3. mood and emotional control: 9 items, 4. communication and understanding: 7 items, 5.daily activities: 10 items, 6. mobility at home and community: 9 items, 7. hand function: 5 items, 8. participation in life: 8 items.
  each item should be rated on on 5-point Lickert scale with 1= extremely difficult OR can't do at all OR no strength at all OR all the time AND 5 means: a lot of strength OR not difficult at all OR none of the time OR Question 9 regarding "recovery from stroke" rated on a scale from 0 - 100 (0= no recovery, 100= full recovery)
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Technology Arm
Number analyzed (Participants) | 14
units on a scale
  pre-intervention | 50 (35)
  post-intervention | 65.5 (17.5)

4. Secondary Outcome: Box and Block Test
Description: Measures broader motoric function of the arm and hand as a performance test. Subjects are required to grab and sort wooden blocks from one side of a small dividing wall set up on a table in front of the sitting subject to another side.
  The unit of the measure is the amount of blocks transferred within 60 seconds.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: blocks/60 sec
Arm/Group | Technology Arm
Number analyzed (Participants) | 14
blocks/60 sec
  pre-intervention | 0 (19.8)
  post-intervention | 1 (30.8)

5. Secondary Outcome: Functional Ambulation Categories (FAC)
Description: Observer based measurement to rate the ability to walk independently. Rated from 0 to 6 (0= not able to walk independently, 6= can walk independently in every situation)
Time Frame: Baseline and 4 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Technology Arm
Number analyzed (Participants) | 14
units on a scale
  pre-intervention | 2 [0 to 5]
  post-intervention | 3.5 [1 to 5]

6. Secondary Outcome: 10m Walk Test= TMT Comfortable
Description: time needed to walk 10 m with Comfortable walking speed
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Technology Arm
Number analyzed (Participants) | 12
seconds
  pre-intervention | 28.6 (22.9)
  post-intervention | 19.0 (19.6)

7. Secondary Outcome: Walking Index of the Chedoke-McMaster Stroke Assessment Measure (CMSA)
Description: The Walking Index consists of the 5 following items:
  Walking indoors Walking outdoors, over rough ground, ramps, and curbs Walking outdoors several blocks Stairs Age and sex appropriate walking distance in meters for 2 minutes
  scored on a 7-point scale (Stage 1 through 7, most impairment through to no impairment, respectively) score from 5 to 35 points, the more points the better
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Technology Arm
Number analyzed (Participants) | 14
units on a scale
  pre-intervention | 16 (8.3)
  post-intervention | 19 (7.8)

8. Secondary Outcome: Berg Balance Scale (BBS)
Description: Observer based measurement of walking, standing and balance with 14 items/task to perform by the subject and rated each on scale from 0 to 4 (0= not able to do without help, 4 = can do safely and independently) score between 0 to 56, the more the better
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Technology Arm
Number analyzed (Participants) | 14
units on a scale
  pre-intervention | 32 (24)
  post-intervention | 39 (18.8)

ADVERSE EVENTS:
Time Frame: over the 4 weeks rehabilitation period
Arm/Group | Technology Arm
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT03641651/Prot_SAP_001.pdf